CLINICAL TRIAL: NCT07158463
Title: Experience With Therapeutic Plasma Exchange in the Pediatric Nephrology Unit of Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shohanda Ahmed Mohamed, Resident of pediatrics, Sohag University
Other Study IDs: Soh-Med--25-8-7MS
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Experience With Therapeutic Plasma Exchange in the Pediatric Nephrology Unit

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Plasmapheresis also known as a therapeutic plasma exchange (TPE) TPE is an extracorporeal blood purification technique designed for the removal of large-molecular-weight substances. Examples of these substances include pathogenic autoantibodies, immune complexes, cryoglobulins, myeloma light chains, endotoxin, and cholesterol-containing lipoproteins Document the indications, procedures, outcomes, and complications associated with TPE in pediatric patients at Sohag University Hospital.

To compare our findings with existing national and international data to identify areas for improvement and standardization.

To evaluate the safety and efficacy of TPE in our pediatric nephrology unit.

ELIGIBILITY:
Inclusion Criteria:

All pediatric patients (aged 1-18 years) who underwent TPE during the study period.

Both male and female.

Exclusion Criteria:

Patients who cannot tolerate central line placement Patients who are in an actively septic state or are hemodynamically unstable . Patients who have allergies to fresh frozen plasma (FFP) or albumin, depending on the type of plasma exchange

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients (aged 1-18 years) who underwent TPE during the study period.
  Both male and female.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of therapeutic plasma exchange in pediatric nephrology unit | One month after last session

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided